CLINICAL TRIAL: NCT06573840
Title: A Functional MRI Study: Assessing Brain Function in Post Stoke Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: business re-focus
Sponsor: NeuroGlove LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REG-1005
Record Dates: First submitted 2023-11-03; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Stroke; Stroke; Acute Ischemic Stroke
Keywords: Stroke; Ischemic Stroke; Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: 3 healthy volunteers and 10 post stroke patients will be enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Cohort (Healthy Cohort) (Active Comparator): Healthy participants who participate in 1 study visit. The unhealthy participant will undergo one functional MRI before, during and after a NeuroGlove session.
  Interventions: Device: NeuroGlove
- Treatment Arm (Active Comparator): The treatment cohort which consists of patients who have experienced an acute ischemic stroke will participate in 1 study visit. They will undergo 1 function MRI before, during and after a NeuroGlove session.
  Interventions: Device: NeuroGlove

INTERVENTIONS:
Device: NeuroGlove — NeuroGlove is a non-invasive device that provides peripheral somatosensory stimulation to the hand. NeuroGlove provides sensory stimulation in the form of pneumatic puffs of air.

SUMMARY:
This is a prospective, single center, observational clinical study containing two cohorts the healthy cohort and post stroke cohort. A total of 13 subjects will be enrolled. Three (3) healthy volunteers will be enrolled in the healthy cohort. Ten (10) subjects who have recently experienced a mild to moderate acute ischemic stroke will be enrolled in the post stroke cohort.

DETAILED DESCRIPTION:
This is a prospective, single center, observational clinical study containing two cohorts the healthy cohort and post stroke cohort. A total of 13 subjects will be enrolled. Three (3) healthy volunteers will be enrolled in the healthy cohort. Ten (10) subjects who have recently experienced a mild to moderate acute ischemic stroke will be enrolled in the post stroke cohort.

Up to13 subjects will be enrolled and complete study procedures. There will be 2 study cohorts enrolled in the study:

1. Healthy Cohort: 3 healthy volunteers (enrolled from the general population)
2. Post Stroke Cohort: 10 subjects who have experienced mild to moderate stroke symptoms that did not completely resolve after acute interventions. (Mild to moderate stroke symptoms is defined as a NIHSS score of 5 to 15.)

ELIGIBILITY:
Inclusion Criteria (Healthy Cohort):

Able and willing to provide informed consent. Men and women ≥18 and <85 years of age. Subject must be right hand dominant. Subject should not have any physical limitations of either upper extremity (e.g., fracture, joint deformity, severe spasticity/contracture, wounds, skin breakdown, lymphedema, etc.)

Inclusion Criteria (Treatment Cohort):

Able to and willing to provide informed consent. Legally authorized representatives (LARs) will not be allowed to consent on behalf of the subject.

Men and women ≥18 and <85 years of age. First single acute ischemic stroke with an onset date within 14 days (± 7 days from onset) of enrollment (time of informed consent) into the study.

Mild to moderate acute ischemic stroke defined as NIHSS score of 3 to 15. Measurable weakness of one upper extremity without complete paralysis (detectable movement in at least 3 fingers).

Subject must be right hand dominant. Subject should not have any physical limitations of either upper extremity (e.g., fracture, joint deformity, severe spasticity/contracture, wounds, skin breakdown, lymphedema, etc.)

Exclusion Criteria:

Coma, inability to cooperate with the study based on impaired level of consciousness or confusion.

Known neurological deficit prior to stroke (including but not limited to previous stroke, MS, Parkinson's disease).

Physical limitations of the weak upper extremity (e.g., fracture, joint deformity, severe spasticity/contracture, wounds, skin breakdown, lymphedema, etc.) Any contraindication to the imaging required per the protocol. Complete middle cerebral artery infarction based on imaging. Carotid artery stenosis >50% of the normal diameter segment (diameter stenosis, compared to the angiographically normal proximal or distal segment).

Subjects has a known history of substance abuse (drug) or alcohol dependence, or lacks the ability to comprehend or following instructions, or for any reason, in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements.

If female, subject is pregnant at the time of enrollment or planning to become pregnant during the trial period.

Subject has any other acute or chronic condition that the investigator believes will adversely affect the ability to interpret the data or will prevent the subject from completing the trial procedures.

Currently participating in another interventional clinical trial. (Observational clinical trial participation is allowed for study enrollment.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Brain Function | 2 hours
  Evaluate brain function through a functional MRI (fMRI) in both healthy subjects (without history of stroke) and post stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Nussbaum, MD, Study Director — NeuroGlove LLC

IPD SHARING:
Plan to Share IPD: No